CLINICAL TRIAL: NCT06111651
Title: Family-Based Prevention to Promote the Social-Emotional Functioning and Healthy Lifestyle Behaviors of Black & Latinx Children
Brief Title: Family-Based Prevention With Black and Latinx Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Daniel Cooper, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00124236; 5P20GM130420 (NIH)
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Child Behavior; Health Behavior
Keywords: parent training; randomized controlled trial; pilot study; child development; implementation trial; prevention
MeSH Terms: conditions — Child Behavior; Health Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): parents will participate in a multicomponent parenting intervention
  Interventions: Behavioral: Parenting Intervention
- Control (No Intervention): parents will receive information about healthy eating habits

INTERVENTIONS:
Behavioral: Parenting Intervention — parent training program with an added emphasis on ethnic-racial socialization and healthy lifestyle behaviors
  Arms: Intervention

SUMMARY:
The main objective of this project is to test whether providing parenting support, with an added emphasis on ethnic-racial socialization and healthy lifestyle behaviors, improves the social-emotional functioning and healthy lifestyle behaviors of Black and Latinx children.

DETAILED DESCRIPTION:
This pilot project is novel in that it (a) interweaves positive parenting practices, ethnic-racial socialization, and healthy lifestyle behaviors into a prevention program for Black and Latinx families, and (b) targets preschool-aged children using a brief, universal prevention approach, which increases potential for dissemination and scalability. The guiding hypothesis is that incorporating these components into a parenting intervention will lead to improvements in children's health as compared to a control condition. A type 1 hybrid effectiveness-implementation design is used to simultaneously test intervention effectiveness while also gathering information on intervention delivery to inform future implementation trials. The specific aims are to: (a) test the preliminary effects of a preventive intervention on the social-emotional functioning and healthy lifestyle behaviors of Black and Latinx children, (b) identify the preliminary effects of the intervention on parenting outcomes, and (c) examine potential barriers and facilitators to intervention delivery.

ELIGIBILITY:
Inclusion Criteria:

Eligible children will:

* be between the ages of 3-6 years
* identify as Black/African American or Latinx/Hispanic
* have a parent or caregiver willing to participate in the intervention that: (a) lives in the same household as the child ≥50% of the time, (b) has primary responsibility for the child, and (c) speaks English or Spanish.

Exclusion Criteria:

Consistent with typical methods associated with a universal prevention approach, there are minimal exclusion criteria. Children will be excluded who:

* have a cognitive/psychological condition that limits the child's ability to communicate
* have a physical health condition that limits the child's ability to be physically active

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2026-01-21 (Actual)

PRIMARY OUTCOMES:
child social-emotional functioning | pre (weeks 0-2) and post intervention (weeks 6-8)
  Parent-reported assessment of various positive and negative child behaviors. Likert scale values range from 0 to 2, with higher values typically indicating greater dysfunctional behavior.
child physical activity | pre (weeks 0-2) and post intervention (weeks 6-8)
  Time spent sedentary and in light, moderate, and vigorous physical activity each day will be collected using a waterproof accelerometer. Validated methods will be used to identify valid days and derive activity intensities.
child sleep | pre (weeks 0-2) and post intervention (weeks 6-8)
  Child average nightly sleep duration and quality will be calculated from data obtained using a waterproof accelerometer.

SECONDARY OUTCOMES:
parenting practices | pre (weeks 0-2) and post intervention (weeks 6-8)
  Parent-reported measure of different dimensions of parenting (e.g., harsh parenting, permissive parenting). Likert scale values range from 1 to 7, with higher values indicating greater dysfunctional parenting.
ethnic-racial socialization practices | pre (weeks 0-2) and post intervention (weeks 6-8)
  Parent-reported measure of attitudes about and use of various ethnic-racial socialization practices. Likert scale values range from 1 to 5, with higher values indicating more positive ethnic-racial socialization attitudes and practices.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States